CLINICAL TRIAL: NCT03465501
Title: Interstitial Brachytherapy Boost for Treatment of Anal Canal Cancers, Comparison of Two Dose Rates
Acronym: BOOST-CA
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BOOST-CA IPC 2017-016
Record Dates: First submitted 2018-03-05; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Anal Canal Cancer
Keywords: Anal Canal Cancer; brachytherapy
MeSH Terms: conditions — Anal Canal Carcinoma | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Dose Rate: Patients treated with brachytherapy at low dose rate of the anal canal with aim of boost
  Interventions: Radiation: Brachytherapy
- High Dose Rate: Patients treated by brachytherapy with a high dose rate of the anal canal aiming for boost
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — Brachytherapy

SUMMARY:
Comparative retrospective study of two anal canal brachytherapy techniques aimed at boosting [low dose rate (LDR) and high dose rate (HDR)]

DETAILED DESCRIPTION:
Efficacy of anal canal interstitial brachytherapy evaluated by local relapse rate, Tolerance of interstitial brachytherapy of the anal canal evaluated by the rate of chronic toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by brachytherapy anal canal to boost.

Exclusion Criteria:

* Patients below age of 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with anal canal brachytherapy for boost, between 2008 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-08-17 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of interstitial brachytherapy of the anal canal | 1 year
  Efficacy of anal canal interstitial brachytherapy evaluated by local relapse rate
Evaluation of the tolerance of interstitial brachytherapy of the anal canal | 1 year
  Tolerance of interstitial brachytherapy of the anal canal evaluated by the rate of chronic toxicities.

SECONDARY OUTCOMES:
Estimation of local control | 1 year
  Local control defined as the time between the date of diagnosis and the date of local relapse or death or recent news
Estimation of disease free survival | 1 year
  Disease free survival defined as the delay between the date of diagnosis and the date of local or locoregional or distant relapse or death or recent news
Estimation of overall survival | 1 year
  Overall survival defined as the time between the date of diagnosis and the date of death or latest news
Comparison of the incidence of toxicities (CTCAE v4) between the 2 groups | 1 year
  rate of toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Leonel VARELA GAGETTI, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordoba A, Escande A, Leroy T, Mirabel X, Coche-Dequeant B, Lartigau E. Low-dose-rate interstitial brachytherapy boost for the treatment of anal canal cancers. Brachytherapy. 2017 Jan-Feb;16(1):230-235. doi: 10.1016/j.brachy.2016.07.007. Epub 2016 Sep 3. PMID 27600606
- [Result] Boukhelif W, Ferri-Molina M, Mazeron R, Maroun P, Duhamel-Oberlander AS, Dumas I, Martinetti F, Guemnie-Tafo A, Chargari C, Haie-Meder C. Interstitial pulsed-dose-rate brachytherapy for the treatment of squamous cell anal carcinoma: A retrospective single institution analysis. Brachytherapy. 2015 Jul-Aug;14(4):549-53. doi: 10.1016/j.brachy.2015.03.006. Epub 2015 Apr 29. PMID 25935731